CLINICAL TRIAL: NCT02205762
Title: LCH-IV, International Collaborative Treatment Protocol for Children and Adolescents With Langerhans Cell Histiocytosis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: North American Consortium for Histiocytosis (Other)
Collaborators: Histiocyte Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-428; 2011-001699-20 (EudraCT Number); 042011 (Other: Children's Cancer Research Institute)
Record Dates: First submitted 2014-07-07; First posted 2014-07-31 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Langerhans cell histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Prednisone; Vinblastine; Mercaptopurine; Indomethacin; Methotrexate; Cytarabine; Cladribine; Hematopoietic Stem Cell Transplantation; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Stratum I (Experimental): Stratum I The combination of Prednisone and vinblastine is the standard first-line combination for patients needing systemic therapy (Stratum I). Patients with MS-LCH and involvement of risk organs, who do not respond to 6-12 weeks of standard therapy, will be immediately switched to alternative treatment approaches (Stratum III or Stratum IV).
  Further therapy prolongation (12 vs. 24 months) and intensification (± mercaptopurine) will further reduce the reactivation rate and the permanent consequences.
  Interventions: Drug: Prednisone; Drug: Vinblastine; Drug: mercaptopurine
- Stratum II (Experimental): A uniform "intensive" 24-week course consisting of prednisolone, vincristine and cytosine-arabinoside will be introduced in Stratum II for eligible patients. It will be followed by a continuation therapy to total treatment duration of 24 months. Participants who after SL-IT (week 24) have a response (NAD or AD better) are eligible for randomization between the continuation arms "INDOMETHACIN" and "6-MP/MTX" (mercaptopurine and Methotrexate).
  Interventions: Drug: Prednisone; Drug: Vinblastine; Drug: mercaptopurine; Drug: INDOMETHACIN; Drug: Methotrexate; Drug: Cytosine Arabinoside
- Stratum III (Experimental): Salvage treatment for risk LCH To assess the efficacy of the combination 2-CdA/Ara-C (Cytosine Arabinoside and 2-chlorodeoxyadenosine) in MS-LCH (patients with risk organ involvement, who fail to respond to front-line (Stratum I) therapy.
  The initial therapy consists of 2 courses of 2-CdA/Ara-C. Continuation of outlined treatment to be assessed at assigned intervals in each stratum.
  Interventions: Drug: 2-chlorodeoxyadenosine
- Stratum IV (Experimental): To determine the overall and disease free survival at 1 and 3 years after reduced intensity conditioning hematopoietic stem cell transplantation (RIC-HSCT). Salvage treatment option for MS-LCH patients with risk organ involvement, who fail to respond to front-line therapy (Stratum I) OR to the salvage 2- CdA/Ara-C regimen (Stratum III).
  Interventions: Procedure: hematopoietic stem cell transplantation (RIC-HSCT)
- Stratum V (Experimental): Stratum V Monitoring and Treatment of isolated tumorous and neurodegenerative CNS-LCH
  - Special regimens will be offered to patients with isolated tumorous CNS-LCH (repeated 2-CdA courses) and to patients with clinically manifested ND-CNS-LCH (+/- extracranial LCH manifestations). For the last group monotherapy with Ara-C courses or (Intravenous immunoglobulin)IVIG will be offered depending on physician's choice.
  Interventions: Drug: Cytosine Arabinoside; Drug: 2-chlorodeoxyadenosine; Biological: Intravenous immunoglobulin
- Stratum VI (Experimental): Natural history and management of "other" SS-LCH not eligible for stratum I group 2.
  * Treatment Options- Management (mostly "wait & see" and topical treatment) is left to the discretion of the treating physician. All treatments and disease responses must be reported in the database. In the case of uncertainties please contact your National Coordinator.
  * Patients being followed on Stratum VI who have progression of disease to MSLCH, multifocal bone disease or CNS-risk bone lesions should be enrolled on Stratum I therapy.
  * Patients being followed on Stratum VI who develop isolated tumorous or neurodegenerative CNS-LCH should be enrolled on Stratum V.
  Interventions: Drug: Prednisone; Drug: Vinblastine; Drug: mercaptopurine; Drug: Cytosine Arabinoside; Drug: 2-chlorodeoxyadenosine; Biological: Intravenous immunoglobulin

INTERVENTIONS:
Drug: Prednisone — Stratum I
  Arms: Stratum I; Stratum II; Stratum VI
Drug: Vinblastine — Stratum I
  Other Names: Velban®; Vincaleukoblastine Sulfate
  Arms: Stratum I; Stratum II; Stratum VI
Drug: mercaptopurine — Stratum I
  Other Names: -Purinethol®; -6-MP
  Arms: Stratum I; Stratum II; Stratum VI
Drug: INDOMETHACIN — Indomethacin fixed dose given daily orally in two divided doses with gastric protection for total treatment duration of 24 months.
  Arms: Stratum II
Drug: Methotrexate — fixed dose weekly orally for total treatment duration of 24 months.
  Arms: Stratum II
Drug: Cytosine Arabinoside
  Other Names: Cytarabine, Ara-C
  Arms: Stratum II; Stratum V; Stratum VI
Drug: 2-chlorodeoxyadenosine
  Other Names: 2-CdA; Cladribin®; Leustatin®
  Arms: Stratum III; Stratum V; Stratum VI
Procedure: hematopoietic stem cell transplantation (RIC-HSCT)
  Arms: Stratum IV
Biological: Intravenous immunoglobulin
  Other Names: IVIG
  Arms: Stratum V; Stratum VI

SUMMARY:
The LCH-IV is an international, multicenter, prospective clinical study for pediatric Langerhans Cell Histiocytosis LCH (age < 18 years).

DETAILED DESCRIPTION:
The international efforts of the past 20 years have shown that combination therapy with vinblastine and prednisone is an effective therapy for Multi-system (MS)-LCH. The previous prospective trial LCH-III confirmed this regimen as a standard regimen for MS-LCH in patients with and without risk organ involvement. It also showed that prolonged treatment in the latter group (treatment duration of 12 vs. 6 months) is superior in preventing disease reactivations. The results of this trial are encouraging and serve as a basis for the LCH-IV study design.Due to the complexity of the disease presentations and outcomes, the LCH-IV study seeks to tailor treatment based on features at presentation and on response to treatment, leading to seven strata:

* Stratum I: First-line treatment for MS-LCH patients (Group 1) and patients with Single system (SS)-LCH with multifocal bone or "Central Nervous System (CNS)-risk" lesions (Group 2)
* Stratum II: Second-line treatment for non-risk patients (patients without risk organ involvement who fail first-line therapy or have a reactivation after completion of first-line therapy)
* Stratum III: Salvage treatment for risk LCH (patients with dysfunction of risk organs who fail first-line therapy)
* Stratum IV: Stem cell transplantation for risk LCH (patients with dysfunction of risk organs who fail first-line therapy)
* Stratum V: Monitoring and treatment of isolated tumorous and neurodegenerative CNS-LCH
* Stratum VI: Natural history and management of "other" SS-LCH (patients who do not need systemic therapy at the time of diagnosis)
* Stratum VII: Long-term Follow up (all patients irrespective of previous therapy will be followed for reactivation or permanent consequences once complete disease resolution has been achieved and the respective protocol treatment completed)

ELIGIBILITY:
Inclusion Criteria:

* Stratum I

  * Patients must be less than 18 years of age at the time of diagnosis.
  * Patients must have histological verification of the diagnosis of Langerhans cell histiocytosis according to the criteria described in Section 6.1
  * Signed informed consent form
* Stratum II

  * Patients of Stratum I who have:
  * Progressive disease (AD worse) in non-risk organs after 6 weeks (Initial Course
  * AD intermediate or worse in non-risk organs or AD better in risk organs after 12 weeks (Initial Course 2)
  * Disease progression (AD worse) in non-risk organs at any time during continuation treatment
  * Active disease at the end of Stratum I treatment
  * Disease reactivation in non-risk organs at any time after completion of Stratum I treatment
* Stratum III

  * Patients from Stratum I who fulfill the following criteria:
  * AD worse in risk organs after week 6 (after Initial Course 1), or AD worse or AD intermediate in risk organs after week 12 (after Initial Course 2).
  * Presence of unequivocally severe organ dysfunction at the above mentioned evaluation points (hematological dysfunction, liver dysfunction, or both of them) as

    * Hb <70 g/L (<7.0 g/dl) and/or transfusion dependency
    * PLT <20 x109/L (20,000/μL) and/or transfusion dependency (both criteria have to be fulfilled) AND/OR
    * Liver dysfunction (or digestive involvement with protein loss)
    * Total protein <55 g/L or substitution dependency
    * Albumin <25 g/L or substitution dependency (at least one of the two criteria to be fulfilled)
* Stratum IV

  * Patients from Stratum I or Stratum III who fulfill the following criteria:
  * AD worse in risk organs after week 6 (after Initial Course 1), or AD worse or AD intermediate in risk organs after week 12 (after Initial Course 2) of Stratum I OR
  * AD worse after the 2nd and 3rd 2-CdA/Ara-C course, and those AD worse or AD intermediate after the 4th 2-CdA/Ara-C course of Stratum III AND
  * Presence of unequivocally severe organ dysfunction at the above mentioned evaluation points (hematological dysfunction, liver dysfunction, or both of them) as defined in Table XI (see Section 10.3.1).
  * Informed consent: All patients or their legal guardians (if the patient is <18 years of age) must sign an Ethics or institutional Review Board approved consent form indicating their awareness of the investigational nature and the risks of this study. When appropriate, younger patients will be included in all discussions in order to obtain assent.
  * Adequate organ function: Patients should have adequate hepatic, renal, cardiac and pulmonary function to undergo reduced intensity HCT based upon local institutional guidelines, or at a minimum meet requirements noted in eligibility checklist Appendix A-VIII_1. However, significant hepatic and pulmonary dysfunction, if secondary to underlying LCH disease activity, will not exclude patients from protocol enrollment and should be discussed with the National PI Coordinator and the Coordinating Principal Investigator.
* Stratum V

  * All patients with verified diagnosis of LCH and MRI findings consistent with ND-CNSLCH irrespective of previous treatments (also those not registered to other Strata ofLCH-IV).
  * Patients with isolated tumorous CNS-LCH (including isolated DI with mass lesion in the hypothalamus-pituitary axis). In patients with already established diagnosis of LCH and radiologic finding of CNS lesions compatible with LCH, a biopsy of the lesion is not obligatory. In all other cases a biopsy of the lesion is needed for inclusion into the study
* Stratum VI

  -- Patients with newly diagnosed SS-LCH and localization other than "multifocal bone",isolated tumorous CNS lesion, or isolated "CNS-risk" lesion.
* Stratum VII -- All patients registered in LCH IV (regardless of treatment) as long as consent for longterm follow-up has not been withheld.

Exclusion Criteria:

* Stratum I

  * Pregnancy (patients of child-bearing age must be appropriately tested before chemotherapy)
  * LCH-related permanent consequences (e.g. vertebra plana, sclerosing cholangitis, lung fibrosis, etc.) in the absence of active disease
  * Prior systemic therapy
* Stratum II

  * Patients with progressive disease in risk organs
  * Permanent consequences (e.g. sclerosing cholangitis, lung fibrosis, etc.) without evidence of active LCH in the same organ or in any other locations
  * No written consent of the patient or his/her parents or legal guardian
* Stratum III

  * The presence of any of the following criteria will exclude the patient from the study:
  * Isolated sclerosing cholangitis without evidence of active hepatic LCH as the only evidence of risk organ involvement.
  * Inadequate renal function as defined by serum creatinine > 3x normal for age
* Stratum IV

  * Pulmonary failure (requiring mechanical ventilation) not due to active LCH.
  * Isolated liver sclerosis or pulmonary fibrosis, without active LCH.
  * Uncontrolled active life-threatening infection.
  * Decreased renal function with a GFR of less than 50ml/1.73m2/min.
  * Pregnancy or active breast feeding
  * Failure to provide signed informed consent
* Stratum VI

  * Patients with SS-LCH who have an isolated tumorous CNS lesion (they are eligible for Stratum V),
  * Patients with isolated "CNS-risk" or multifocal bone lesions (they are eligible for Stratum I, Group 2)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2016-11-02; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with Reactivation Free Survival | 12 Months
  Stratum I, II, VI
Response Rate of Second Cycle | 9 weeks
  Stratum III
Overall and disease free survival at 1 and 3 years after reduced intensity conditioning hematopoietic stem cell transplantation (RIC-HSCT) | 3 Years
  Stratum IV
The cumulative incidence of radiological and clinical neurodegeneration in patients with isolated tumorous CNS-LCH, DI, anterior pituitary dysfunction, and those with CNS-risk lesions | 2 Years
  Stratum V
The time interval and cumulative incidence of progression of radiological neurodegeneration to clinically manifested ND-CNS-LCH | 2 Years
  Stratum V
Cumulative incidence of specific Permanent Consequences e.g. diabetes insipidus (DI), growth hormone deficiency (GHD), neuropsychological impairment, etc. | 2 Years
  From all treatment stratum via long-term follow up in Stratum VII

SECONDARY OUTCOMES:
Overall Survival | 2 Years
  Stratum I
Number of Participants with Serious and Non-Serious Adverse Events | 2 Years
Incidence of Permanent Consequences | 2 Years
  All Stratum
Cumulative incidence of reactivations in risk organs | 2 Years
Time to complete disease resolution | 2 Years
  Stratum III
Response rate to the combination of prednisone, vincristine and cytarabine | 2 years
  Stratum II
The proportion of patients alive and free of disease without permanent consequences (e.g. diabetes insipidus, anterior pituitary dysfunction, radiological or clinical neurodegeneration) | 2 Years
  Stratum II
Percentage of treatment-related toxicities | 2 Years
  Stratum II
Reactivation rates after continuation treatment with Indomethacin vs. 6-MP/MTX. | 2 years
  Stratum II
The type of subsequent intensive and/or maintenance therapy utilized | 2 Years
  Stratum III
Early and late mortality | 2 Years
  Stratum II
Early and late toxicity | 2 Years
  Stratum III
d+100 transplant related mortality | 2 Years
  Stratum IV
Incidence of hematopoietic recovery, and donor chimerism at d+100 and 1 year post RIC-HSCT | 2 Years
Record all occurrence of skin, GI or liver abnormalities fulfilling criteria of Grades II-IV acute GVHD | 2 Years
  Stratum IV: Hematopoetic Stem Cell Transplantation for Risk LCH
Percentage of Participants with incidence of chronic GVHD | 2 Years
  Stratum IV
Response Rate to ND-CNS-targeted therapy at 12 and 24 months after start of therapy | 2 years
  Stratum V
Response of isolated tumorous CNS-LCH to 2-CDA | 2 Years
  Stratum V
Frequency of ND-CNS-LCH in patients with isolated tumorous CNS-LCH | 2 Years
  Stratum V
Methods of early identification of ND-CNS-LCH | 2 Years
  Stratum V - Exploration of the value of neurochemistry, neurophysiology, and neuropsychology methods in early identification of ND-CNS-LCH and in assessing its severity, and comparison to MRI findings.
Need for systemic therapy later during disease course | 2 Years
  Stratum VI
Identify possible risk factors for permanent consequences (PC) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Milen Minkov, MD, Ph.D, Study Chair — Children's Cancer Research Institute / St. Anna Children's Hospital; Carlos Rodriguez-Galindo, MD, Study Chair — North American Consortium for Histiocytosis
Locations (42):
- United States (42):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Valley Children's Healthcare, Madera, California
  - UCSF Benioff Children's Hospital of Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Helen Diller Family Cancer Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Emory, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Children's Mercy Hospitals, Kansas City, Kansas
  - University of Kentucky A.B.Chandler Medical Center, Lexington, Kentucky
  - University of Louisville, Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Minnesota, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University / Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Carolinas Medical Center, Levine Children's Hospital, Charlotte, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, University Hospitals, Cleveland, Ohio
  - Russell J Ebeid Children's Hospital (Promedica), Toledo, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Greenville Health System BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Children's Medical Center Dallas, UT Southwestern, Dallas, Texas
  - Providence Sacred Heart Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - American Family Children's Hospital University of Wisconsin, Madison, Wisconsin